CLINICAL TRIAL: NCT03128320
Title: A Randomized, Single-blind, Threefold Crossover, Single-center Study to Assess the Safety and the Effects of 1 mg and 5 mg BAY1193397 in Comparison to Placebo on Skin Capillary Blood Flow and Transcutaneous Oxygen Pressure After Single Dose in Type II Diabetic Patients
Brief Title: The Effects of BAY1193397 on Skin Capillary Blood Flow and Transcutaneous Oxygen Pressure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 17500; 2015-003799-63 (EudraCT Number)
Record Dates: First submitted 2017-04-21; First posted 2017-04-25 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Diabetic Foot
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BAY1193397/Placebo (sequence A-B-C) (Experimental): Subjects with type II diabetes who follow treatment sequence A-B-C. Single oral dose of a placebo tablet in the first intervention period (Treatment A); followed by single oral dose of 1 mg BAY1193397 (Treatment B); then single oral dose of 5 mg BAY1193397 IR tablet under fasted state in the third intervention period (Treatment C). A wash-out phase of approximately 120 - 360 hours was maintained between each treatment.
  Interventions: Drug: BAY1193397; Drug: Placebo
- BAY1193397/Placebo (sequence B-C-A) (Experimental): Subjects with type II diabetes who follow treatment sequence B-C-A. Single oral dose of 1 mg BAY1193397 in the first intervention period (Treatment B); followed by single oral dose of 5 mg BAY1193397 IR tablet under fasted state in the second intervention period (Treatment C), then single oral dose of a placebo tablet under fasted conditions in the third intervention period (Treatment A). A wash-out phase of approximately 120 - 360 hours was maintained between each treatment.
  Interventions: Drug: BAY1193397; Drug: Placebo
- BAY1193397/Placebo (sequence B-A-C) (Experimental): Subjects with type II diabetes who follow treatment sequence B-A-C. Single oral dose of 1 mg BAY1193397 in the first intervention period (Treatment B); followed by single oral dose of a placebo tablet in the second intervention period (Treatment A), then 5 mg BAY1193397 IR tablet under fasted conditions in the third intervention period (Treatment C). A wash-out phase of approximately 120 - 360 hours was maintained between each treatment.
  Interventions: Drug: BAY1193397; Drug: Placebo

INTERVENTIONS:
Drug: BAY1193397 — Single dose of 1 mg BAY1193397 given in the fasted state
Drug: BAY1193397 — Single dose of 5 mg BAY1193397 given in the fasted state
Drug: Placebo — Single dose of placebo given in the fasted state

SUMMARY:
The purpose of the study is to analyse skin blood flow in diabetic patients. The patients receive a single dose of placebo, 1 mg BAY1193397, and 5 mg BAY1193397. The analysis of safety and tolerability are secondary objectives of this study.

ELIGIBILITY:
Inclusion Criteria:

* The informed consent must be signed before any study specific tests or procedures are done (patient must be able to give informed consent, no legal representative allowed)
* Patients with a diagnosis of type II diabetes mellitus and PAD (peripheral artery disease) and/or microangiopathy as evidenced by at least one of the following criteria:

  1. TBPI (toe / brachial blood pressure index) < 0.7 at screening
  2. ischemic or neuro-ischemic DFU (diabetic food ulcer) in medical history (verified by medical records)
  3. clinical diagnosis of PAD in medical history (verified by medical records)
  4. diagnosis of nephropathy that is most likely due to diabetes mellitus type II
  5. diagnosis of diabetic retinopathy
  6. diagnosis of diabetic polyneuropathy
* Age 55 to 75 years (inclusive) at the screening visit
* Non-smokers are preferred for inclusion in this study. If smokers are included, they must refrain from smoking on the days of treatment periods 1, 2, and 3 until all examinations have been performed
* Patients are expected to be on stable medication during study conduct. No planned changes in drug therapy during active treatment period of the study (i.e. from treatment period 1 to treatment period 3) is allowed.
* Men or confirmed postmenopausal women (defined as exhibiting spontaneous amenorrhea for at least 12 months before screening or as exhibiting spontaneous amenorrhea for 6 months before screening with documented serum follicle-stimulating hormone [FSH] levels > 40 mIU/mL) or women without childbearing potential based on surgical treatment 6 weeks before screening such as bilateral tubal ligation, bilateral oophorectomy with or without hysterectomy (documented by medical report verification). Male patients, who are sexually active and have not been surgically sterilized must agree to use two reliable and acceptable methods of contraception simultaneously (one method used by the study patient and one method used by the partner) during the study and for 12 weeks after receiving the investigational medicinal product and not to act as sperm donor for 12 weeks after dosing. Acceptable methods of contraception include for example: a) condoms (male or female) with or without a spermicidal agent b) diaphragm or cervical cap with spermicide c) intrauterine device d) hormone-based contraception
* Ability to understand and follow study related instructions

Exclusion Criteria:

* Patients with existing lower limb ulcers
* Patients with nailfold capillaries at the great toe that are technically difficult to assess
* Patients suffering from PAD Fontaine Stage 4
* Patients requiring planned revascularization
* Patients suffering from diseases other than diabetes mellitus that are known to lead to disturbances in skin microcirculation or interfering with the method of measurement such as Raynaud's disease, collagen vascular disorders , atopic dermatitis, psoriasis
* Myocardial infarction, acute coronary syndrome, transient ischemic attack (TIA), stroke, revascularization, angioplasty within 3 months prior to randomization
* Any planned surgical intervention during the course of the study
* Medical condition or history thereof or any deviation from normal laboratory values that in the opinion of the investigator would impair the ability to complete the planned study procedures.
* Any surgical or medical condition which significantly alters absorption, distribution, metabolism or excretion of study drugs, including, but not limited to: history of major gastrointestinal (GI) tract surgery, inflammatory bowel disease, currently active gastritis, pancreatitis, treatment with cholestyramine and colestipol resins
* Patients with HbA1c > 12% (> 108 mmol/mol) at the screening visit
* Any other condition or therapy, which would make the subject unsuitable for this study and will not allow participation for the full planned study period (e.g. active malignancy or other condition limiting life expectancy to less than 12 months)
* Use of alpha- or beta-AR (adrenoreceptor) agonists
* Use of alpha-AR antagonists
* Use of serotonin/norepinephrine reuptake inhibitors (SNRIs)
* Use of tricyclic antidepressants at a dose equivalent of more than 50 mg amitryptyline
* No pedicure or nail polish is allowed from screening until the end of the active study period (end of treatment period 3)
* Systolic blood pressure below 100 mmHg or above 180 mmHg at the screening visit based on the average of three readings taken from the arm with the highest systolic recordings
* Diastolic blood pressure below 50 or above 110 mmHg at the screening visit based on the average of three readings taken from the arm with the highest systolic recordings
* Heart rate below 50 or above 100 beats/min at screening (obtained from ECG)
* Clinically relevant findings in the physical examination which, in the opinion of the investigator, preclude participation for reasons of the patient's safety
* Estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73m^2 using the Modification of Diet in Renal Disease (MDRD) formula at screening

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-05-25 (Actual); Primary Completion 2019-09-06 (Actual); Study Completion 2019-10-28 (Actual)

PRIMARY OUTCOMES:
Change in resting capillary blood flow velocity (CBV) | Before and after treatment with study drug (within 1-3 hours after treatment with study drug)
  = resting CBV after study drug administration - resting CBV before study drug administration
Change in peak CBV during reactive hyperemia | Before and after treatment with study drug (within 1-3 hours after treatment with study drug)
  = peak CBV after study drug administration - peak CBV before study drug administration
Change in time to peak CBV during reactive hyperemia | Before and after treatment with study drug (within 1-3 hours after treatment with study drug)
  = time to peak CBV after study drug administration - time to peak CBV before study drug administration
Change in transcutaneous oxygen pressure (TcPO2) | Before and after treatment with study drug (within 1-3 hours after treatment with study drug)
  = TcPO2 after study drug administration - TcPO2 before study drug administration

SECONDARY OUTCOMES:
Number of subjects with treatment-emergent adverse events (TEAEs) | From first application of study medication up to 2 days after end of treatment with study medication
Number of subjects with TEAEs in different severity | From first application of study medication up to 2 days after end of treatment with study medication

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Royal Devon & Exeter Hospital, Exeter, Devon, United Kingdom

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/